CLINICAL TRIAL: NCT04410744
Title: Incidence and Risk Factors for Trocar Site Incisional Hernia Detected by Clinical and Ultrasonographic Examination.
Brief Title: Incidence and Risk Factors for TSIH
Acronym: TSIHi
Status: Completed | Type: Observational
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Ana Ciscar, General and digestive surgery specialist, Hospital de Mataró
Other Study IDs: TSIH INCIDENCE
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Incisional Hernia
Keywords: Incisional hernia; Port site; Trocar site; Risk factors; Incidence
MeSH Terms: conditions — Incisional Hernia | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonographic examination — All clinical examinations (physical exam) and ultrasounds are performed by a single surgeon and a single radiology resident supervised by the same abdominal radiology consultant, respectively.
  Other Names: Clinical examination

SUMMARY:
Trocar site incisional hernia (TSIH) is the most frequent complication associated to laparoscopic surgery. Few studies currently describes its real prevalence or risk factors. The aim of this study is to determine the real incidence of TSIH and to identify risk factors in the investigator's series of patients.

A cross sectional, prospective study is performed including consecutive patients who underwent a laparoscopic procedure during a four months period. All the patients are assessed both clinically (TSIHc) and by an ultrasonographic exam (TSIHu). Main variable studied is the incidence of TSIH. A multivariate analysis is performed to identify risk factors.

DETAILED DESCRIPTION:
Single-centre cross-sectional study based on prospective clinical and radiological assessment and retrospective risk factor analyses performed at a single hospital.

All consecutive patients who underwent laparoscopic surgery (cholecystectomy, colon resection, adrenalectomy, Nissen fundoplication and appendectomy) during a four months period were included in the study. At least 30 months after hospital discharge, they were invited by telephone to participate in the study. Detailed project information was provided, and those who accepted received an appointment for an outpatient visit and a dynamic ultrasound. Informed consent was obtained from all participants. In all patients, the umbilical trocar wound was closed with an interrupted suture with synthetic braided absorbable 2/0 suture (Novosyn® or Safil®). During the postoperative outpatient visit, clinical and ultrasonographic examinations were performed. To increase study homogeneity, all clinical examinations and ultrasounds were performed by a single surgeon and a single radiology resident supervised by the same abdominal radiology consultant, respectively. Sonography was performed with an Applio 500 equipment (Toshiba, Japan) with a 3.5MHz convex probe and a 7MHz linear probe. The ultrasound diagnosis was based on the identification of an abdominal wall defect with intraabdominal tissue protrusion. The main variables of the study were clinical (TSIHc) and ultrasound (TSIHu) diagnosis of incisional hernia. All results and variables were introduced in a previous specifically designed database (File MakerPro 11.0v3 © 1984-2011 FileMaker, Inc.). Data were collected from clinical interviews, physical and radiological examinations and the electronic medical record. Statistical analyses were performed using the SPSS statistical software (IBM SPSS® Statistics).

ELIGIBILITY:
Inclusion Criteria:

* Previous laparoscopic surgery
* Age ≥18 years
* Informed consent signed

Exclusion Criteria:

* Previous umbilical hernia repair
* Age < 18 years
* Informed consent not signed
* Failure to attend the postoperative appointment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who underwent laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
clinical TSIH incidence | 30 seconds
  Presence / absence palpableTSIH (yes / not)
ultrasonographic TSIH incidence | 1 minute 30 seconds
  Identification of an abdominal wall defect with intraabdominal tissue protrusion (yes /not) Caudal and cranial diameters of the abdominal wall's defect (cm)

SECONDARY OUTCOMES:
Risk factors for TSIH | 5 minutes
  Risk factors for TSIH determination. Information obtained from the electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ciscar, Principal Investigator — Hospital de Mataró

REFERENCES:
- [Derived] Ciscar A, Badia JM, Novell F, Bolivar S, Mans E. Incidence and risk factors for trocar-site incisional hernia detected by clinical and ultrasound examination: a prospective observational study. BMC Surg. 2020 Dec 14;20(1):330. doi: 10.1186/s12893-020-01000-6. PMID 33317503